CLINICAL TRIAL: NCT06963216
Title: A Phase III Open-Label Multi-Center Study of the Pharmacokinetics, Safety, and Efficacy of Coagadex in the Treatment of Adults With Acquired Factor X Deficiency Associated With Light Chain Amyloidosis
Brief Title: A Study Investigating Coagadex in the Treatment AFXD Associated With AL Amyloidosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kedrion S.p.A. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB074; IRAS UK # 1011593 (Other: United Kingdom Health Research Authority)
Record Dates: First submitted 2025-04-14; First posted 2025-05-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Acquired Factor X Deficiency
Keywords: Factor X Deficiency; Blood Coagulation Disorders; Hematologic Diseases; Hemorrhagic Disorders; Light Chain amyloidosis; AL amyloidosis
MeSH Terms: conditions — Factor X Deficiency; Blood Coagulation Disorders; Hematologic Diseases; Hemorrhagic Disorders; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Masking Description: None (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- On-Demand Treatment Cohort (Experimental): Participants without an active bleeding event will enter the Run-In Period, which lasts up to 180 days. Upon a bleeding event participants will receive a first dose of 40 IU/kg of Coagadex®. Additional dose(s) will be based on the incremental recovery (IR). (If an allowed Emergent Surgery becomes necessary in the Run-In Period, the participant will cross over into the Surgery/Invasive Procedures Cohort.)
  Interventions: Biological: Coagadex(R)
- Surgery/Invasive Procedures Cohort (Experimental): Participants enrolled at least 3 weeks prior to a scheduled surgical intervention will undergo pharmacokinetic sampling. The dose of Coagadex® will be determined based on the patient's PK profile. (During this 3-week period, if the participant develops an acute bleed, they will cross over into the On-Demand Treatment Cohort for treatment.)
  Interventions: Biological: Coagadex(R)

INTERVENTIONS:
Biological: Coagadex(R) — Coagulation Factor X (Human)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Coagadex in treating active bleeds and to manage peri-operative bleeding in participants with acquired factor X deficiency associated with AL amyloidosis.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of Coagadex® in treating active bleeds and to manage peri-operative bleeding in participants with aFXD associated with AL amyloidosis. Coagadex® is a plasma-derived human coagulation factor concentrate expected to treat bleeding episodes in patients with aFXD associated with AL amyloidosis by delivering concentrated Factor X to address the clotting deficiency caused by the disease.

aFXD is a rare condition (prevalence of <1 / 1 000 000 [Orphanet 2024]) and may occur due to infections, neoplastic and chronic diseases (Lee G et al., 2012). aFXD is considered severe when the FX coagulant activity (FX:C) level is < 25% of normal (normal range 70 - 150 IU/dL), and moderate when FX:C level is 25% to 50% of normal (Choufani et al., 2001).

AL amyloidosis is the most common cause of acquired FX Deficiency (aFXD). In AL amyloidosis, amyloid fibrils bind to and reduce the levels of circulating FX and shorten its half-life, causing aFXD, leading to an increase in risk of bleeding. Bleeding may occur both in patients with moderate and severe deficiency

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ages 18-70 years old.
2. Diagnosis of aFXD associated with AL amyloidosis with FX:C ≤ 50 IU/dL.
3. Woman of Childbearing Potential (defined in Appendix 2) and men of reproductive potential who agree to use an effective contraception measure during the study.

Exclusion Criteria:

1. Female participants that are pregnant or lactating.
2. Presence of FX inhibitors.
3. Uncontrolled arterial hypertension.
4. On anticoagulant therapy (not antiplatelets), unstable heart disease, clinically significant thrombotic event in the past 180 days or any other condition that the Investigator believes is likely to interfere with evaluation of the study drug or with satisfactory conduct of the trial.
5. Any factor X containing product taken within 2 weeks of first Coagadex® administration.
6. Participation in another interventional clinical study with an investigational drug, biologic, or device within 30 days prior to screening.
7. Hemodynamically unstable due to any cause or even after blood transfusion, fluid resuscitation and pharmacologic or volume replacement pressor therapy.
8. Prior history of bleeding disorder other than aFXD.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of bleeding events responsive to Coagdex® therapy at 72 hours after initiation of treatment in the On-Demand Treatment Cohort | at 72 hours
  Proportion of bleeding events with a 'positive' response.
Proportion of bleeding events responsive to Coagdex® therapy at 72 hours after initiation of treatment in the Surgery/Invasive Procedures Cohort | at 72 hours
  Proportion of bleeding events with a 'fair, good, or excellent' response.

SECONDARY OUTCOMES:
Proportion of bleeding events responsive to Coagdex® therapy at Different Timepoints After 72 hours in the On- Demand Cohort | Day 4 to day 30
  Investigators will assess Coagadex® efficacy in the on-demand treatment cohort by looking at: -Percentage of responsive bleedings, -The ability to discontinue or reduce the dose and/or dosing frequency of Coagadex®.
To assess the safety of Coagadex® by number and percentage of infusion related AEs, SAEs, coded by MedDRA | Day 0 through study completion, an average of up to 6 months.
  To assess the safety of Coagadex® in the on-demand treatment of bleeding and management of peri-operative/peri-procedural hemostasis in infusion related AEs and SAEs. AEs and SAEs will be evaluated following the first Coagadex® administration: assessment of seriousness, causality assessment; and incidence, frequency, and severity of AEs and incidence and frequency of SAEs.
Proportion of bleeding events responsive to Coagdex® therapy at Different Timepoints After 72 hours in Surgery/Invasive Procedures Cohort | Day 4 to Day 14
  Investigators will assess Coagadex® efficacy in the surgery/invasive procedures cohort by looking at:
  * The overall percentage of bleeding episodes successfully controlled,
  * The ability to discontinue or reduce the dose and/or dosing frequency of Coagadex®.
Coagadex® exposure | Day 1 to Day 30
  Assess the number of study drug exposure days (overall and per participant) and the Coagadex® exposure per event.
Assess Post-treatment FX Levels | Day 1 to Day 30
  Assess in the on-demand treatment cohort and surgery/invasive procedures cohort by FX:C IU/mL
Assess bleeds at other sites. | Last Coagadex® until study completion, an average of up to 6 months.
  Description: Assessed in the surgery/invasive procedures cohort by looking at: Number of sites per participant including severity, duration, location, and cause.
Assess the pharmacokinetics(PK) of Coagadex® in peri-operative/peri-procedural hemostasis in Surgery/Invasive Procedures Cohort. | Day 0 pre-dose to Day 5
  To assess the pharmacokinetics(PK) of Coagadex® in peri-operative/peri-procedural hemostasis by PK parameter Maximum Plasma Concentration [Cmax]

CONTACTS AND LOCATIONS:
Overall Officials: Mirella Calcinai, MD, Study Director — Medical Director, Clinical Development
Locations (2):
- United States (2):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No
Publishing of data and IPD that underlie results in the publication will be determined at study completion to comply with ICMJE minimum requirements.